CLINICAL TRIAL: NCT02362373
Title: Women With Epilepsy: a Pilot Study of Pharmacokinetic and Pharmacodynamic Anti-epileptic Drug Effects in Levonorgestrel Intrauterine System Users
Brief Title: Women With Epilepsy: a Pilot Study of PK and PD Anti-epileptic Drug Effects in Levonorgestrel Intrauterine System Users
Acronym: WESAIL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Anne Davis, Associate Professor of Clinical Obstetrics and Gynecology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AAAI0750
Record Dates: First submitted 2015-02-09; First posted 2015-02-12 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2015-12

CONDITIONS: Epilepsy; Contraception
Keywords: epilepsy; contraception; drug interaction
MeSH Terms: conditions — Epilepsy | interventions — Levonorgestrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- levonorgestrel IUS (Other): all women in the study underwent placement of the levonorgestrel IUS in an open-label fashion, outcomes were compared before and after placement.
  Interventions: Drug: levonorgestrel IUS

INTERVENTIONS:
Drug: levonorgestrel IUS — placement of levonorgestrel intrauterine system
  Other Names: Mirena

SUMMARY:
The investigators will conduct a prospective, seven-month pilot study to explore pharmacokinetic (PK) and pharmacodynamic (PD) effects among women with epilepsy using the levonorgestrel intrauterine system (LNG IUS) for contraception. The investigators will enroll twenty women with well-controlled epilepsy maintained on stable anti-epileptic drugs (AED) therapy seeking the LNG IUS for contraception. The primary outcomes are AED levels and seizures before and after LNG IUS placement. Secondary outcomes include LNG levels, evidence of ovulation three weeks after insertion (serum progesterone >3ng/ml), bleeding and spotting, endometrial thickness, continuation, satisfaction and adverse events (removals, expulsions, side effects). The investigators will conduct a baseline month assessment, insertion visit, and follow-up visits at 21 days, three months and six months.

DETAILED DESCRIPTION:
Study Procedures This pilot study consists of five study visits. Once preliminary eligibility is determined through a telephone screening interview, the first visit is scheduled.

Visit 1 Enrollment/Baseline

* Review Eligibility
* Informed Consent
* Collect Baseline Information
* Vital Signs
* Pregnancy Test
* Complete Physical Exam including Pelvic exam,
* Chlamydia testing, and a Pap test if needed as per ASCCP (American Society for Colposcopy and Cervical Pathology) guidelines
* Receive diary to record any bleeding or spotting
* Receive condoms, if needed, for use until IUS insertion
* Sign release for contact of primary neurologist or epileptologist
* Study MD to contact participant's neurologist to notify of trial participation, and verify type and dose of AEDs

Visit 2 Insertion/4-6 Weeks from Baseline

* Vital Signs
* Pregnancy Test
* Phlebotomy for hormone and AED levels
* Transvaginal ultrasound
* IUS Insertion
* Review and collect completed diary
* Receive new diary

Visit 3/ Follow up 3 Weeks post IUS Insertion

* Vital Signs
* Phlebotomy for hormone and AED levels
* Transvaginal Ultrasound
* Review and collect completed diary
* Receive new diary

Visit 4/Follow up 3 Months post IUS Insertion

* Vital Signs
* Phlebotomy for hormone and AED levels
* Transvaginal ultrasound
* Review and collect completed diary
* Receive new diary
* Acceptability Questionnaire

Visit 5/ Exit 6 Months post IUS insertion

* Vital Signs
* Phlebotomy for hormone and AED levels
* Transvaginal Ultrasound
* Review and collect final completed diary
* Acceptability Questionnaire

ELIGIBILITY:
Inclusion Criteria:

1. Age18-45 years
2. Regular menstrual cycle of length 21-35 days
3. Willing to use IUS for contraception
4. Willing to use non-hormonal contraception for one month before insertion
5. Stable AED therapy for at least two months
6. Well-controlled epilepsy (2 or fewer seizures, other than simple partial, per month)
7. Working telephone
8. English Speaking

Exclusion Criteria:

1. Current pregnancy or pregnancy in the previous two months
2. Breastfeeding with amenorrhea
3. Hepatic p450 enzyme inducing medications other than AEDs (griseofulvin, rifampin, St. John's Wort, bosentan)
4. Depomedroxyprogesterone acetate within previous six months
5. Congenital or acquired uterine anomaly, including myomas, that distort the uterine cavity
6. Acute pelvic infection or a history pelvic infection without subsequent intrauterine pregnancy
7. Postpartum endometritis or infected abortion in the last three months
8. Genital bleeding of unknown etiology
9. Untreated lower genital tract infection (cervical or vaginal)
10. Acute liver disease or liver tumor, benign or malignant
11. HIV infection or partner with HIV infection
12. Increased susceptibility to pelvic infection
13. A previously inserted intrauterine device (IUD) that has not been removed
14. Hypersensitivity to any component of the LNG IUS
15. Known or suspected carcinoma of the breast
16. Current abnormal cervical cytology other than ASCUS or a history of abnormal cervical cytology other than ASCUS without appropriate follow-up demonstrating no evidence of disease
17. History of genital tract malignancy
18. Current use of anti-coagulants
19. Current alcoholism or drug abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Davis, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Derived] Vieira CS, Pack A, Roberts K, Davis AR. A pilot study of levonorgestrel concentrations and bleeding patterns in women with epilepsy using a levonorgestrel IUD and treated with antiepileptic drugs. Contraception. 2019 Apr;99(4):251-255. doi: 10.1016/j.contraception.2018.11.018. Epub 2018 Dec 4. PMID 30529085

RESULTS

PARTICIPANT FLOW:
Groups:
- Women With Epilepsy Receiving the LNG IUS: There was one group in this pilot study. All women received the LNG IUS.
Period: Overall Study
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Levonorgestrel IUS
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants That Experienced Clinically Meaningful Change in Lamotrigine Level
Description: The outcome measure is designed to examine whether participants will experience subtherapeutic or toxic serum trough level of lamotrigine after IUD insertion.
Time Frame: from baseline to 6 months after LNG IUS insertion
Population: 13 out of 20 participants received lamotrigine while on IUD.
Measure: Number; unit: percentage of participants
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Number analyzed (Participants) | 13
percentage of participants | 0

2. Primary Outcome: Percent of Participants That Experienced Clinically Meaningful Change in Levetiracetam Level
Description: The outcome measure is designed to examine whether participants will experience subtherapeutic or toxic serum trough level of levetiracetam after IUD insertion.
Time Frame: from baseline to 6 months after LNG IUS insertion
Population: 5 out of 20 participants received levetiracetam while on IUD.
Measure: Number; unit: percentage of participants
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Number analyzed (Participants) | 5
percentage of participants | 0

3. Primary Outcome: Percent of Participants That Experienced Clinically Meaningful Change in Oxcarbazepine Level
Description: The outcome measure is designed to examine whether participants will experience subtherapeutic or toxic serum trough level of oxcarbazepine after IUD insertion.
Time Frame: from baseline to 6 months after LNG IUS insertion
Population: 3 out of 20 participants received oxcarbazepine while on IUD.
Measure: Number; unit: percentage of participants
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Number analyzed (Participants) | 3
percentage of participants | 0

4. Secondary Outcome: Change in Seizure Frequency
Description: Number of participants with increased, unchanged or decreased mean monthly seizure frequency.
Time Frame: baseline to 6 months
Measure: Number; unit: participants
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Number analyzed (Participants) | 20
participants
  Seizure control unchanged | 13
  Seizure control decreased | 3
  Seizure control improved | 4

5. Secondary Outcome: Number of Participants Continuing With IUD
Description: Women continuing the IUD for contraception at 6 months
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Number analyzed (Participants) | 20
participants | 20

ADVERSE EVENTS:
Arm/Group | Women With Epilepsy Receiving the LNG IUS
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 5/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women With Epilepsy Receiving the LNG IUS (N=20)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2) — One participant had a cyst that ruptured; conservative management was successful and no surgery was required.
Uterine cramping (Reproductive system and breast disorders) | 5 (5)
urinary tract infection (Renal and urinary disorders) | 2 (2)
Stomach pain (Gastrointestinal disorders) | 2 (2)
Muscle spasms (General disorders) | 2 (2)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
acne (Skin and subcutaneous tissue disorders) | 1 (1)
common cold (General disorders) | 1 (1)
vaginal itching (Reproductive system and breast disorders) | 2 (2)
flu (General disorders) | 1 (1)
yeast infection (Reproductive system and breast disorders) | 1 (1)
hemmorhoids (Gastrointestinal disorders) | 1 (1)
sinus congestion (General disorders) | 2 (2)
bacterial vaginosis (Reproductive system and breast disorders) | 2 (2)
palpitations (Cardiac disorders) | 1 (1)
bladder spasms (Renal and urinary disorders) | 1 (1)
hip injury (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (Nervous system disorders) | 1 (1)
herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
shoulder surgery (Musculoskeletal and connective tissue disorders) | 1 (1)
pelvic pain (Reproductive system and breast disorders) | 1 (1)
seasonal allergies (General disorders) | 1 (1)
pinched nerve (Nervous system disorders) | 1 (1)
strep throat (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes